CLINICAL TRIAL: NCT06097728
Title: A Phase III, Randomized, Open-Label, Multicenter, Global Study of Volrustomig (MEDI5752) in Combination With Carboplatin Plus Pemetrexed Versus Platinum Plus Pemetrexed or Nivolumab Plus Ipilimumab in Participants With Unresectable Pleural Mesothelioma (eVOLVE-Meso)
Brief Title: MEDI5752 in Combination With Carboplatin Plus Pemetrexed in Unresectable Pleural Mesothelioma
Acronym: eVOLVE-Meso
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D7988C00001; 2023-503231-17-00 (Registry Identifier: CTIS (EU)); 2023-000067-32 (EudraCT Number)
Record Dates: First submitted 2023-10-04; First posted 2023-10-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Unresectable Pleural Mesothelioma
Keywords: Mesothelioma; Pleural Mesothelioma; Unresectable Pleural Mesothelioma; Advanced pleural mesothelioma
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant | interventions — Pemetrexed; Carboplatin; Cisplatin; Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: This is a randomized, open-label, Phase III trial in participants with untreated unresectable pleural mesothelioma. Approximately 825 participants across histology subtypes will be randomized in a 1:1 ratio to receive volrustomig in combination with carboplatin plus pemetrexed or the investigator's choice of nivolumab plus ipilimumab or platinum plus pemetrexed chemotherapy for participants with epithelioid histology, and nivolumab plus ipilumab for participants with non-epithelioid histology.
Who Masked: Outcomes Assessor
Masking Description: This is an open-label study for the personnel at study sites; the specific treatment to be taken by a participant will be assigned using an Interactive Response Technology/Randomization and Trial Supply Management. To maintain the integrity of the study, AstraZeneca personnel directly involved in the study conduct will not undertake or have access to efficacy data aggregated by treatment arm prior to final data readout for the primary endpoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Volrustomig + Carboplatin + pemetrexed (Experimental): Volrustomig in combination with carboplatin plus pemetrexed
  Interventions: Drug: Volrustomig; Drug: Pemetrexed; Drug: Carboplatin
- Investigator's choice of standard care (Active Comparator): The investigator's choice of nivolumab plus ipilimumab or platinum plus pemetrexed chemotherapy for participants with epithelioid histology, and nivolumab plus ipilumab for participants with non-epithelioid histology.
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Volrustomig — MEDI5752: Administered as IV infusion
  Other Names: MEDI5752
  Arms: Volrustomig + Carboplatin + pemetrexed
Drug: Pemetrexed — Alimta: Administered as IV infusion
  Other Names: Alimta
Drug: Carboplatin — Paraplatin: Administered as IV infusion
  Other Names: Paraplatin
Drug: Cisplatin — Platinol: Administered as IV infusion
  Other Names: Platinol
  Arms: Investigator's choice of standard care
Drug: Nivolumab — Opdivo: Administered as IV infusion
  Other Names: Opdivo
  Arms: Investigator's choice of standard care
Drug: Ipilimumab — Yervoy: Administered as IV infusion
  Other Names: Yervoy
  Arms: Investigator's choice of standard care

SUMMARY:
This is a phase III, randomized, open-label, multicenter, global study to determine the efficacy and safety of Volrustomig (MEDI5752) + Carboplatin + Pemetrexed vs the investigator's choice of platinum + Pemetrexed or Nivolumab + Ipilimumab in participants with unresectable pleural mesothelioma.

DETAILED DESCRIPTION:
Adult patients with histologically proven diagnosis of pleural mesothelioma with advanced unresectable disease are eligible to be enrolled. Patients will be randomized 1:1 to receive Volrustomig (MEDI5752) + Carboplatin + Pemetrexed or the investigator's choice of platinum+Pemetrexed or Nivolumab+Ipilimumab, based on their histology.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant must be ≥ 18 years at the time of screening
* Histologically proven diagnosis of pleural mesothelioma with known histology (epithelioid vs. non-epithelioid)
* Advanced unresectable disease that cannot be treated with curative surgery (with or without chemotherapy)
* WHO/ECOG performance status of 0 or 1 with no deterioration (that is, ECOG PS>1) over the previous 2 weeks prior to day of first dosing
* Has measurable disease per modified RECIST1.1
* Has adequate bone marrow reserve and organ function at baseline

Key Exclusion Criteria:

* As judged by the investigator, any condition that would interfere with evaluation of the investigational product or interpretation of participant safety or study results.
* Active or prior documented autoimmune or inflammatory disorders
* History of another primary malignancy with exceptions.
* Uncontrolled intercurrent illness
* Tuberculosis, hepatitis B (HBV) or hepatitis C (HCV), human immunodeficiency virus (HIV) infection that is not well controlled
* Any concurrent chemotherapy, radiotherapy, investigational, biologic, or hormonal therapy for cancer treatment
* Untreated or progressive CNS metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2027-11-19 (Estimated); Study Completion 2028-11-16 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) in experimental arm relative to comparator arm | up to approximately 61 months
  OS is defined as the time from randomization until the date of death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to approximately 61 months
  OS is defined as the time from randomization until the date of death due to any cause.
Progression Free Survival (PFS) | up to approximately 61 months
  PFS is defined as the time from randomization until progression per mRECIST 1.1 and/or RECIST 1.1 as assessed by the investigator at local site, or death due to any cause.
Landmark OS | 12, 18, 24, 36 months
  Landmarks of OS12, OS18, OS24, and OS36.
Landmark PFS | 6, 12, 18, 24 months
  Landmarks of PFS6, PFS12, PFS18, and PFS24
Overall Response Rate (ORR) | up to approximately 61 months
  Proportion of participants who have a confirmed Complete Response or confirmed Partial Response, as determined by the investigator at local site per mRECIST 1.1 and/or RECIST 1.1.
Duration of Response (DoR) | up to approximately 61 months
  DoR defined as the time from the date of first documented response until date of documented progression per mRECIST 1.1 and/or RECIST 1.1 as assessed by the investigator at local site or death due to any cause.
PFS2 | up to approximately 61 months
  PFS2 defined as the time from randomization to the earliest of the progression event (following the initial investigator-assessed progression), after first subsequent therapy, or death.
Patient-reported physical functioning | up to approximately 61 months.
  TTD in physical functioning as measured by PROMIS (Patient Reported Outcomes Measurement Information System) Physical Function Short Form 8c. There are 8 questions each from a scale of 1 (unable to do) to a scale of 5 (With a little difficulty). The higher the scores the better the patient-reported physical functioning is.
Disease-related symptoms using EORTC IL305 (Q1) | Up to approximately 61 months.
  Change from baseline in disease-related symptoms as measured by individual symptom items from the EORTC (European Organisation For Research And Treatment Of Cancer) IL305 (Item Library 305) (Q1). It is scored from a 1 (not at all) to a 4 (very much). The higher the score the higher the disease-related symptoms.
Disease-related symptoms using PRO-CTCAE (Q1, 5, 6, 9) | Up to approximately 61 months
  Change from baseline in disease-related symptoms as measured by individual symptom items from the PRO-CTCAE (Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events) (Q1, 5, 6, 9). PRO-CTCAE responses are scored from 0 to 4 (or 0/1 for absent/present). The higher the score the higher the disease-related symptoms.
Patient-reported role functioning using EORTC QLQ-C30 RF subscale (IL305 Q2 3) | up to approximately 61 months
  Change from baseline in functioning will be assessed by the following measure:
  Role functioning: EORTC (European Organisation For Research And Treatment Of Cancer) QLQ (Quality of Life Questionnaire) -C30 RF (Role Functioning) subscale (IL305 Q2 3) (Item Library 305). The questions are from a scale of 1 (not at all) to 4 (very much). The lower the score the higher the patient-reported role functioning is.
Patient-reported HRQoL (Health-related Quality of Life) using EORTC QLQ-C30 HRQoL subscale (IL305 Q7-8) | Up to approximately 61 months
  Change from baseline in functioning will be assessed by the following measure:
  HRQoL: EORTC (European Organisation For Research And Treatment Of Cancer) QLQ (Quality of Life Questionnaire) -C30 HRQoL subscale (IL305 Q7-8) (Item Library 305). The questions are from a scale of 1 (very poor) to 7 (excellent). The higher the score the higher the HRQoL.
Immunogenicity of volrustomig | up to approximately 61 months
  Incidence of Anti-Drug Antibodies against volrustomig.
Incidence of Adverse Events (AEs) AEs graded by CTCAE version 5.0 | Up to approximately 61 months
  Incidence of Adverse Events (AEs) AEs graded by CTCAE (Common Terminology Criteria for Adverse Events) version 5.0. Grade refers to the severity of the AE. The CTCAE displays grade 1 (mild) through 5 (death related to AE). Grade 2 (moderate), Grade 3 (Severe) and Grade 4 (Life-threatening consequences).
Area under the curve (AUC) | Up to approximately 61 months
  The concentration of MEDI5752 in serum will be determined. Area under the curve is the integral of the concentration-time curve. The AUC reflects the actual body exposure to drug after administration. The AUC is dependent on the rate of elimination of the drug from the body and the dose administered.
Maximum plasma concentration of the drug (Cmax) | Up to approximately 61 months
  The concentration of MEDI5752 in serum will be determined (Cmax will be derived).
The time taken to reach the maximum concentration (Tmax) | Up to approximately 61 months
  The concentration of MEDI5752 in serum will be determined (Tmax will be derived).

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie G Zauderer, MD, Principal Investigator — Memorial Slone Kettering (MSK) Cancer Centre; Arnaud Scherpereel, MD, Principal Investigator — Lille University
Locations (161):
- United States (20):
  - Research Site, Phoenix, Arizona
  - Research Site, Duarte, California
  - Research Site, Santa Rosa, California
  - Research Site, Aurora, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, East Brunswick, New Jersey
  - Research Site, Commack, New York
  - Research Site, Valhalla, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Independence, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
- Australia (5):
  - Research Site, Chermside
  - Research Site, Clayton
  - Research Site, Melbourne
  - Research Site, Nedlands
  - Research Site, Westmead
- Belgium (6):
  - Research Site, Anderlecht
  - Research Site, Antwerp
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Leuven
  - Research Site, Sint-Niklaas
- Brazil (7):
  - Research Site, Barretos
  - Research Site, Fortaleza
  - Research Site, João Pessoa
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santo André
  - Research Site, São Paulo
- Canada (7):
  - Research Site, Edmonton, Alberta
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- China (21):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Ningbo
  - Research Site, Qingdao
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- Denmark (2):
  - Research Site, Aarhus N
  - Research Site, Copenhagen
- France (12):
  - Research Site, Brest
  - Research Site, Créteil
  - Research Site, Le Mans
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Rouen
  - Research Site, Saint-Herblain
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (12):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Cologne
  - Research Site, Essen
  - Research Site, Gauting
  - Research Site, Georgsmarienhütte
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Kiel
  - Research Site, Münster
  - Research Site, Regensburg
- Italy (10):
  - Research Site, Alessandria
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Rozzano
  - Research Site, Varese
- Japan (12):
  - Research Site, Amagasaki-shi
  - Research Site, Hakodate-shi
  - Research Site, Hiroshima
  - Research Site, Kitaadachi-gun
  - Research Site, Kitakyushu-shi
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Nishinomiya-shi
  - Research Site, Okayama
  - Research Site, Osakasayama-shi
  - Research Site, Tokyo
  - Research Site, Ube-shi
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Eindhoven
  - Research Site, Rotterdam
- Norway (2):
  - Research Site, Lørenskog
  - Research Site, Oslo
- Poland (6):
  - Research Site, Bydgoszcz
  - Research Site, Bystra
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Warsaw
- South Africa (6):
  - Research Site, Cape Town
  - Research Site, eManzimtoti
  - Research Site, Johannesburg
  - Research Site, Kimberly
  - Research Site, Polokwane
  - Research Site, Pretoria
- South Korea (3):
  - Research Site, Cheongju-si
  - Research Site, Seoul
  - Research Site, Ulsan
- Spain (4):
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Oviedo
- Switzerland (5):
  - Research Site, Baden
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Fribourg
  - Research Site, Sankt Gallen
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (4):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Diyarbakır
  - Research Site, Izmir
- United Kingdom (9):
  - Research Site, Cambridge
  - Research Site, Cardiff, Wales
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Portsmouth
  - Research Site, Taunton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/